CLINICAL TRIAL: NCT06801288
Title: Diagnostic Role of Renal Biopsy in Patients With Fabry Disease
Acronym: FABRY-SS-21
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: FABRY-SS-21
Record Dates: First submitted 2024-12-30; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, single-centre, non-pharmacological observational study carried out for scientific and health protection purposes. It provides for the systematic collection of information from the medical records of patients with a genetic diagnosis of Fabry Disease referred to the single centre of Renal Genetic Diseases of the IRCCS Azienda Ospedaliero-Universitaria di Bologna.

These patients were considered eligible for the biopsy procedure if:

* presence of a clinical picture compatible with a classical phenotype
* presence of laboratory (microalbuminuria, proteinuria, GFR reduction by various methods) or instrumental (renal ecostructural features) pathological alterations suggestive of Fabry disease
* presence of VUS
* presence of an abnormal course of nephropathy or doubtful overlapping pathology.

Patients with ESRD were excluded.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the diagnostic capacity, currently undocumented in the literature, of renal biopsy in patients with Anderson-Fabry disease, afferent to the Sant'Orsola-Malpighi General Hospital's Single Centre for Renal Genetic Diseases.

As secondary objectives we intend to assess whether the renal damage associated with Fabry disease, evidenced by histological features obtained by biopsy, manifests differently in subgroups of patients defined by:

* Gender
* CKD stage
* genetic mutations Individual pathological lesions are assessed using the Scoring System devised by the International Study Group of Fabry Nephropathy (ISGFN).

All patients with a definite diagnosis of Fabry's disease who have been admitted to the IRCCS Azienda Ospedaliero-Universitaria di Bologna's single centre for Renal Genetic Diseases from 01/01/2012 to 31/12/2020 are eligible. Based on the number of patients afferent to the genetic kidney disease outpatient clinic, approximately 80 patients will be enrolled. The comparison will be performed on the basis of variables that are associated with Fabry disease in the literature, such as enzyme activity assessment, Lyso-GB3 assay, renal function parameters, enzyme therapy, genetic mutations and cardiac markers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age with a diagnosis of Fabry disease defined based on the 2017 guidelines.
* Obtaining written Informed Consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a definite diagnosis of Fabry's disease who have been admitted to the IRCCS Azienda Ospedaliero-Universitaria di Bologna's single centre for Renal Genetic Diseases from 01/01/2012 to 31/12/2020 are eligible. Based on the number of patients afferent to the genetic kidney disease outpatient clinic, approximately 80 patients will be enrolled. The comparison will be performed on the basis of variables that are associated with Fabry disease in the literature, such as enzyme activity assessment, Lyso-GB3 assay, renal function parameters, enzyme therapy, genetic mutations and cardiac markers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic capacity of renal biopsy | Baseline
  The main objective of the study is to evaluate the diagnostic capacity, currently undocumented in the literature, of renal biopsy in patients with Anderson-Fabry disease
Renal damage associated with Fabry disease | Baseline
  To assess whether the renal damage associated with Fabry disease, evidenced by histological features obtained by biopsy, using the Scoring System devised by the International Study Group of Fabry Nephropathy (ISGFN).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Sant'Orsola University Hospital - Nephrology, Dialysis and Transplant Unit, Bologna, BO, Italy